CLINICAL TRIAL: NCT05188326
Title: A Randomized Study to Evaluate the Efficacy of 5-Aza for Post-Remission Therapy of Acute Myeloid Leukemia in Elderly Patients
Brief Title: Efficacy of 5-Aza for Post-Remission Therapy of Acute Myeloid Leukemia (AML) in Elderly Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Associazione Qol-one (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QOLESS-AZA-AMLE
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia,; Post-Remission Therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Injections; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azacitidine (Experimental): Vidaza consists of 50 mg/ m2 s.c or i.v for 7 days (5 + weekend off + 2) every 28 days and increase after 1st cycle, if well tolerated, to 75 mg/m2 s.c or i.v. for 7 days (5 + weekend off + 2) every 28 days for further 5 cycles followed by cycles every 56 days for 4 years and six months
  Interventions: Drug: Vidaza 100 milligram (mg) injection
- Best supportive care (Placebo Comparator): No drug administration
  Interventions: Other: Best Supportive Care

INTERVENTIONS:
Drug: Vidaza 100 milligram (mg) injection — 1st cycle 50 mg/sqm s.c. or i.v. for 7 days (5 + weekend off + 2) every 28 days and increase dosing after 1st cycle, if well tolerated, to 75 mg/ m2 for further 5 cycles, followed by cycles every 56 days for 4 years and six months post-remission.
  Other Names: Vidaza
  Arms: Azacitidine
Other: Best Supportive Care — Best supportive care includes antibiotics, transfusions and fluids
  Arms: Best supportive care

SUMMARY:
The present study aims to compare the efficacy of postremission maintenance therapy with 5-Aza versus best supportive care (BSC) in a cohort of AML patients aged >60 years, who have achieved complete remission (CR) following conventional induction ('3+7') and consolidation chemotherapy.

DETAILED DESCRIPTION:
The present study aims to compare the efficacy of postremission maintenance therapy with 5-Aza versus best supportive care (BSC) in a cohort of AML patients aged >60 years, who have achieved CR following conventional induction ('3+7') and consolidation chemotherapy to evaluate 2 an 5 year post-remission rates of Overall Survival and disease free survival between two arms

ELIGIBILITY:
Inclusion Criteria:

1. Age 61 years or more
2. Newly diagnosed AML with > 30% myeloid marrow blasts, either "de novo" or evolving from a MDS not previously treated with chemotherapeutic agents.
3. Absence of central nervous system involvement
4. No contraindications for intensive chemotherapy, defined as:

   1. prior congestive heart failure requiring treatment and/or left ventricular systolic ejection fraction below the normal range;
   2. a creatinine or bilirubin level more than twice the upper limit of normal, except if AML-related;
   3. a Performance Status (PS) score of > 2;
   4. uncontrolled severe infection.
5. Informed consent.

Exclusion Criteria:

1. Age ≤ 60 years
2. Newly diagnosed AML with < 30% myeloid marrow blasts
3. Previously treated AML
4. Central nervous system involvement
5. Prior congestive heart failure requiring treatment and/or left ventricular systolic ejection fraction below the normal range;
6. A creatinine or bilirubin level more than twice the upper limit of normal, except if AML-related;
7. A PS score of > 2;
8. Uncontrolled severe infection.

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-11-28 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Disease free Survival (DFS) | 5 years
  Disease-free survival (DFS) at 2 and 5 years. Events for DFS are death and first relapse (either AML or myelodysplastic syndrome (MDS) recurrence) and death; observations are censored at the date of last contact if alive and disease-free. DFS will be calculated from the date of achievement of CR to the date of 1st relapse or death. Patients still alive in 1st CR will be censored at the moment of last visit/contact.

SECONDARY OUTCOMES:
Hospitalizations | 5 years
  Number and length of hospitalizations in the post-remission period.
Overall Survival (OS) | 2 and 5 years
  Overall survival (OS) at 2 and 5 years. Event for OS in both arms is death and patients are censored at the date of last contact if alive

CONTACTS AND LOCATIONS:
Overall Officials: Esther Natalie Oliva, Study Chair — QOL-ONE Associazione Culturale e di Ricerca
Locations (18):
- Italy (18):
  - A.O. SS. Antonio e Biagio e Cesare Arrigo, Alessandria, AL
  - Ospedale Riuniti, Ancona, AN
  - A.O. S. Giovanni Moscati, Avellino, AV
  - Policlinico Università di Bari, Bari, BA
  - Ospedale L'Annunziata, Cosenza, CS
  - Ospedale Ferrarotto, Catania, CT
  - Ospedale Garibaldi, Catania, CT
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, FG
  - Università degli Studi di Genova, Genova, GE
  - IRCCS Ospedale Maggiore Policlinico, Milan, MI
  - Ospedale Civile Spirito Santo, Pescara, PE
  - Grande Ospedale Metropolitano Bianchi-Melacrino-Morelli, Reggio Calabria, RC
  - Ospedale Sant'Eugenio, Roma, RM
  - Policlinico Agostino Gemelli, Roma, RM
  - Azienda Ospedaliera Sant'Andrea, Rome, RM
  - IRCCS Istituto Regina Elena, Rome, RM
  - A.O.U. San Giovanni di Dio e Ruggì D'Aragona, Salerno, SA
  - A.O.U. di Udine Centro Trapianti e Terapie Cellulari, Udine

IPD SHARING:
Plan to Share IPD: No